CLINICAL TRIAL: NCT06769048
Title: JADE: Phase II Trial in Patients With Geographic Atrophy: A Randomized, Double-masked, Placebo-controlled, Dose-finding Study to Evaluate the Efficacy and Safety of BI 1584862
Brief Title: A Study to Test Different Doses of BI 1584862 in People With a Distinct Form of Age-related Macular Degeneration (AMD) Called Geographic Atrophy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1484-0005; U1111-1309-9115 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-01-07; First posted 2025-01-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo-matching BI 1584862 (Placebo Comparator)
  Interventions: Drug: Placebo-matching BI 1584862
- BI 1584862 dose 1 (Experimental)
  Interventions: Drug: BI 1584862
- BI 1584862 dose 2 (Experimental)
  Interventions: Drug: BI 1584862
- BI 1584862 dose 3 (Experimental)
  Interventions: Drug: BI 1584862

INTERVENTIONS:
Drug: Placebo-matching BI 1584862 — Placebo-matching BI 1584862
  Arms: Placebo-matching BI 1584862
Drug: BI 1584862 — BI 1584862
  Arms: BI 1584862 dose 1; BI 1584862 dose 2; BI 1584862 dose 3

SUMMARY:
This study is open to adults aged 50 years and older with geographic atrophy that was diagnosed by imaging of the retina. The purpose of this study is to find out whether a medicine called BI 1584862 improves the eyes in people with geographic atrophy and to find the most suitable dose.

This study has 4 treatment groups. Participants are put into groups randomly, which means by chance. Initially participants can join a BI 1584862 and a placebo group; then more participants are put randomly in 2 additional BI 1584862 groups and a placebo group.

Participants are in the study for 1 year. During this time, they visit the study site 13 times. At the visits, doctors check the severity of participants' eye disease and collect information on any health problems. They take detailed pictures of the back of the eye, the retina, with imaging methods called fundus autofluorescence (FAF), near-infrared reflectance (NIR), and optical coherence tomography (OCT). They measure areas of the retina that appear healthy (bright) or start to waste away (dark, atrophy). The changes over time are then compared between the treatment groups.

ELIGIBILITY:
Inclusion criteria:

* Men and women with at least 1 eye with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) determined by fundus autofluorescence (FAF). The total size of all GA lesions in the study eye (as determined by the independent central reading center (CRC)) must be ≥1.25 mm^2 and ≤12.0 mm^2:

  * If multiple lesions are present in the study eye, at least 1 lesion must have an area of ≥0.5 mm^2
  * At least 1 GA lesion must be at least in part within a 1500 μm radius ring centered on the fovea
  * The foveal center point must not be involved in any atrophic lesion
  * Lesion(s) must reside completely within the FAF image
* Best corrected visual acuity (BCVA) score of ≥50 letters in the study eye using the early treatment diabetic retinopathy study (ETDRS) chart (approximately equivalent to ≥20/100 on the Snellen chart).
* Hyperautofluorescence of any pattern, as assessed by the CRC, must be present in the junctional zone of GA in the study eye.
* Age ≥50 years.
* Men must be willing and able to use contraception (condom, abstinence) to prevent pregnancy and/or exposure of an existing embryo or fetus to the investigational product. A female participant is eligible if she is not a woman of childbearing potential.
* Signed informed consent consistent with International Conference of Harmonization-Good Clinical Practice (ICH GCP) guidelines and local legislation

Exclusion criteria:

* Any history of, or evidence of, exudative age-related macular degeneration (eAMD) in the study eye.
* Previously received treatment for GA in the study eye within 4 months or 5 half-lives, prior to baseline, whichever is longer.
* Previously received an investigational medication (oral or intravitreal) for GA within 4 months or 5 half-lives prior to baseline, whichever is longer.
* Additional eye disease in the study eye that could compromise BCVA or significantly impact retinal morphology:

  * uncontrolled glaucoma, defined as a disk-to-cup ratio >0.8 or ocular hypertension with intra ocular pressure (IOP) >24 mmHg at screening visit, or use of >2 active IOP-lowering agents in the study eye
  * clinically significant diabetic retinopathy or maculopathy in the opinion of the investigator
  * history of high myopia, i.e. spherical equivalent of ≥8 diopters or axial length ≥27.2 mm. Note: if subject had prior cataract or refractive surgery, spherical equivalent should be evaluated with pre-operative refraction. If axial length measurement is not available in medical records and cannot be obtained at screening visit, assessment of high myopia can be made by investigator on clinical examination.
  * anterior segment and vitreous abnormalities that would preclude adequate observation with SD-OCT in the opinion of the investigator
  * other ocular conditions at the discretion of the investigator that might interfere with the outcome of the trial
* Significant disease or other medical conditions (as determined by medical history, examination, and clinical investigations at screening) that may, in the opinion of the investigator result in any of the following:

  * put the participant at risk because of participation in the study
  * influence the results of the study
  * cause concern regarding the participant's ability to comply with the protocol requirements or complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the participant an unreliable trial participant)
* Known hypersensitivity to any of the ingredients used in the investigational medicinal product (IMP) formulation, or any of the medications used.
* Active intraocular inflammation in the study eye.
* Active infectious conjunctivitis in either eye. Further exclusion criteria apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
Slope of change from baseline in square root transformed geographic atrophy (GA) area as measured by fundus autofluorescence (FAF) over a treatment period of up to 50 weeks (expressed in mm/year) in the study eye | Up to week 50.
  mm is millimeters.

SECONDARY OUTCOMES:
Key secondary endpoint: Change from baseline in total attenuation as a percentage of the EZ at the macular area with a thickness of 0 μm up to week 50 assessed by volumetric OCT and EZ mapping in the study eye | Up to week 50.
  EZ stands for ellipsoid zone. OCT stands for optical coherence tomography.
Key secondary endpoint: Slope of change from baseline in square root transformed GA area as measured by OCT over a trial period of up to 50 weeks (expressed in mm/year) in the study eye | Up to week 50.
  GA stands for geographic atrophy. OCT stands for optical coherence tomography. mm is millimeters.
Occurrence of TEAES from drug administration until Week 52 | Up to week 52.
Change from baseline in partial attenuation as a percentage of the ellipsoid zone (EZ) at the macular area with thickness <20 micrograms (μm) up to week 50 assessed by volumetric optical coherence tomography (OCT) in the study eye | Up to week 50.
Change from baseline in square root transformed geographic atrophy (GA) area as measured by fundus autofluorescence (FAF) at Week 50 (expressed in mm) in the study eye | At baseline and at week 50.
Occurrence of BCVA letter loss of ≥15 from baseline in the study eye as measured by standardized ETDRS chart for at least 2 consecutive visits between baseline and up to Week 50 | Up to week 50.
  ETDRS is early treatment diabetic retinopathy study.
Change from baseline in best-corrected low luminance visual deficit (LLVD) score as measured in letters by ETDRS chart under low-luminance conditions at Week 50 in the study eye | At baseline and at week 50.
  ETDRS is early treatment diabetic retinopathy study.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (43):
  - Associated Retina Consultants, Gilbert, Arizona
  - Associated Retina Consultants, Ltd., Phoenix, Arizona
  - Cameron Ria, LLC, Phoenix, Arizona
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Global Research Management, Glendale, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Retinal Consultants Medical Group, Inc, Modesto, California
  - Northern California Retina Vitreous Associates MedicalGroup, Inc., Mountain View, California
  - Eye Research Foundation, Newport Beach, California
  - Retina Consultants of San Diego, Poway, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Bay Area Retina Associates - Walnut Creek, Walnut Creek, California
  - Retina Specialists of Colorado Research, LLC, Denver, Colorado
  - Coastal Eye Surgeons, Greenwich, Connecticut
  - Vitreo Retinal Associates - Gainesville, Gainesville, Florida
  - MedEye Associates, Miami, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Illinois Retina Associates - Oak Park, Oak Park, Illinois
  - The Eye Care Institute, Louisville, Kentucky
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - University of Missouri Health System, Columbia, Missouri
  - NJRetina, Teaneck, New Jersey
  - Verum Research, LLC, Eugene, Oregon
  - Retina Northwest, Portland, Oregon
  - EyeHealth Northwest, Portland, Oregon
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Charleston Neuroscience Institute - Charleston, Charleston, South Carolina
  - Tennessee Retina, Nashville, Tennessee
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas-Beaumont-70319, Beaumont, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Red River Research Partners, LLC - Plano, Plano, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Retina Consultants of Texas - Schertz, Schertz, Texas
  - Retina Consultants of Texas-The Woodlands-67575, The Woodlands, Texas
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Pacific Northwest Retina, Bellevue, Washington
- Emanuelli Research & Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency